CLINICAL TRIAL: NCT05238129
Title: Baseline Study on Current Practice of Patients Undergoing C-arm Procedures of Extremities or Spinal Cord at the Operating Department of the Maastricht University Medical Center+
Brief Title: Current Practice of Patients Undergoing C-arm Procedures at the Operating Department
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: NL.MUMC.ORCarms
Record Dates: First submitted 2022-02-03; First posted 2022-02-14 (Actual); Last update posted 2022-04-20 (Actual); Status verified 2022-04

CONDITIONS: Types of C-arm Procedures Included; Low Complex (Lower & Upper Extremities); High Complex (Lower Extremities & Spinal Cord)

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No intervention - standard care is assessed — No intervention - standard care is assessed

SUMMARY:
All x-ray systems at the MUMC+ are currently operated by radiodiagnostic technicians. This is also the case for C-arms used during surgical procedures at the OR-complex. Because a gain in time efficiency is expected (i.e. not for research related reasons), a group of OR-personnel will be in-house trained to qualify for operating C-arms in low complex procedures. The shift towards C-arm procedures performed by OR personnel has been initiated also in other hospitals as it is expected to be time saving without loss of quality. However, this is an assumption and not proven by any scientific evidence. Several aspects are interesting for scientific studies as little is known about the effects of this shift on image quality, radiation dose, time efficiency and to guarantee that there is no loss of quality for the patient.

This study investigates the standard care, where radiodiagnostic technician operate the C-arms.

This study is set up such that it can serve as a baseline for a future study in which it will be assessed whether the quality of care when OR-personnel operates the C-arms is non-inferior to the standard care.

The aim of the study is to prospectively assess the standard care.

Research questions are twofold:

1. What is the current practice and current time efficiency of C-arm procedures performed by radiodiagnostic technicians?
2. What is the current quality of C-arm procedures operated by radiodiagnostic technicians?

ELIGIBILITY:
Inclusion Criteria:

* All C-arm OR-procedures performed at the OR-complex of the MUMC+;
* Type of procedure is: low complex: extremities (upper or lower), high complex: lower extremities, spinal cord (four procedure types).

Exclusion Criteria:

* No informed consent;
* Incomplete procedure information and technical parameters;
* Withdrawal of informed consent by the study patient.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of consecutive patients who undergo a low complex C-arm procedure (lower or upper extremities) or a high complex C-arm procedure (lower extremities or spinal cord) during the study period at the OR complex of the MUMC+.
Sampling Method: Non-Probability Sample
Enrollment: 540 (Estimated)
Dates: Start 2022-05-01 (Estimated); Primary Completion 2023-01 (Estimated); Study Completion 2023-02 (Estimated)

PRIMARY OUTCOMES:
Gross and nett OR time [minutes] | 1 day
  Measures for time efficiency, recorded by assistent investigator during procedure
Radiation dose (DAP[Gycm2]) | 1 day
  Measure for quality

SECONDARY OUTCOMES:
Time spent by and type of personnel involved [minutes, predefined role] | 1 day
  Measure for efficiency, recorded by assistent investigator during procedure
Amount of time spent inefficiently [minutes] | 1 day
  Measure for efficiency, recorded by assistent investigator during procedure
Occupancy time C-arm [minutes] | 1 day
  Measure for efficiency, recorded by assistent investigator during procedure
Downtime (technical failures) [minutes] | 1 day
  Measure for efficiency, recorded by assistent investigator during research period
Number of revision surgeries | 1 month
  Measure for quality, recorded by assistent investigator 1 month after the procedure
Radiation dose (Dose in ref_point [mGy]) | 1 day
  Measure for quality, obtained from C-arm
Image quality subjective scoring | 1 day
  Measure for quality, questionaire, Likert scale 1-5 (5 being highest quality)
Number and type of help requests | 1 day
  Measure of quality and efficiency, recorded by assistent investigator during procedure
Collimation [cm2] | 1 day
  Measure for quality, obtained from the C-arm (= used field size)
Radiation related procedure time (beam on, fluoroscopy and acquisition time) [seconds] | 1 day
  Measure for quality, obtained from the C-arm
Number and types of events | 1 day
  Measure for quality, obtained from the C-arm

IPD SHARING:
Plan to Share IPD: No